CLINICAL TRIAL: NCT02079584
Title: Outpatient Treatment of Low-Risk Venous Thromboembolism With Target Specific Anticoagulant
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: fwa00003543
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Venous Thromboembolism
Keywords: Patient Compliance; Target Specific Anticoagulant; Quality of Life
MeSH Terms: conditions — Venous Thromboembolism; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: None Retained — A blood sample will be obtained at the initial outpatient visit within 30 days (+/- 14 days) post diagnosis and/or start of treatment and at the 180 day (+/- 14 days) follow up post treatment visit and at each annual visit for up to 5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Warfarin: A study group taken from existing anticoagulant clinics treated with warfarin.
- Rivaroxaban: A group seen in the rivaroxaban clinic under study.

SUMMARY:
The objectives of this registry are to measure the outcomes, cost, adherence pattern and experience of patients treated as outpatients with rivaroxaban after being diagnosed with blood clots in the emergency department. The investigators hypothesize that patients will have a relatively low rate of adverse events and higher adherence than has been reported historically for warfarin treatment. Patients will be scheduled for follow up care with one of Dr. Kline's Outpatient Thrombosis clinics at Methodist Hospital, Eskenazi Health Services and the Baylor University Medical Center (Dallas, TX) after diagnosis and treatment of pulmonary embolism (PE) or deep vein thrombosis (DVT).

DETAILED DESCRIPTION:
Information will be obtained from the patient medical records, past medical history, physical examination at initial outpatient clinic visit 30 days (+/- 14 days) and 6 months or 180 days (+/- 14 days) post diagnosis or start of treatment, then annual follow ups for up to 5 years. The data will be collected and stored in a database, the IU RedCap database system will be used to develop a database and store information .

ELIGIBILITY:
Inclusion:

* DVT or PE diagnosed on imaging:
* Systolic always>100 mm Hg in absence of history of low blood pressure
* No contraindication to anticoagulation treatment (active bleeding or high risk postoperative status, creatinine clearance < 30 ml/min, history of heparin induced thrombocytopenia or warfarin skin necrosis);
* No other medical condition requiring hospital treatment (sepsis, new or decompensated existing organ failure, intractable pain);
* No social condition requiring hospital treatment (homelessness with history of non-adherence to treatment, suspected neglect or abuse, incarceration, untreated psychosis, severe alcohol or drug dependency);
* No coagulopathy or current anticoagulant resulting in an INR>1.7, or thrombocytopenia (platelet count < 50,000/uL);
* No need for supplemental oxygen (no respiratory distress and pulse ox always >94%)

Exclusion:

- If active cancer, POMPE-C <6%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Heterogeneous group of patients pulled primarily from an emergency department population, diagnosed with low-risk VTE.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08-14 (Actual); Study Completion 2014-08-14 (Actual)

PRIMARY OUTCOMES:
Clot Recurrence | 5 years
  The primary outcome is clot recurrence, with the rivaroxaban cohort expected to be equivalent or improved with warfarin.
Bleeding | 5 years
  Bleeding that requires change in therapy

SECONDARY OUTCOMES:
Adherence | 5 years
  Number of patients discontinuing anticoagulation in first 30 days and reason why

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beam DM, Kahler ZP, Kline JA. Immediate Discharge and Home Treatment With Rivaroxaban of Low-risk Venous Thromboembolism Diagnosed in Two U.S. Emergency Departments: A One-year Preplanned Analysis. Acad Emerg Med. 2015 Jul;22(7):788-95. doi: 10.1111/acem.12711. Epub 2015 Jun 25. PMID 26113241
- [Background] Kahler ZP, Beam DM, Kline JA. Cost of Treating Venous Thromboembolism With Heparin and Warfarin Versus Home Treatment With Rivaroxaban. Acad Emerg Med. 2015 Jul;22(7):796-802. doi: 10.1111/acem.12713. Epub 2015 Jun 25. PMID 26111453
- [Result] Kline JA, Kahler ZP, Beam DM. Outpatient treatment of low-risk venous thromboembolism with monotherapy oral anticoagulation: patient quality of life outcomes and clinician acceptance. Patient Prefer Adherence. 2016 Apr 15;10:561-9. doi: 10.2147/PPA.S104446. eCollection 2016. PMID 27143861